CLINICAL TRIAL: NCT03437850
Title: Strengthening Health Systems for Persons With Traumatic Spinal Cord Injury in South Africa and Sweden: a Protocol for a Longitudinal Study of Processes and Outcomes
Brief Title: Strengthening Health Systems for Persons With Traumatic Spinal Cord Injury in South Africa and Sweden
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of the Western Cape (Other)
Collaborators: Medical Research Council, South Africa (Other); Karolinska Institutet (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Dr Conran Joseph, Lecturer (PhD), University of the Western Cape
Other Study IDs: BM/16/3/24
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- South African cohort
  Interventions: Other: Usual care
- Swedish Cohort
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Care as usual, in terms of processes and outcomes, will be collected for all participants in both cohorts

SUMMARY:
A traumatic spinal cord injury (TSCI) often causes an unprecedented change in functioning by altering bodily structure and function. More specifically, the direct consequences of TSCI to the motor, sensory and autonomic nervous system not only challenge an individual's independency but also the ability to make a positive adjustment to life after injury. In line with this, TSCI survivors often experience threats to their livelihood and becoming integrated members of society. Health systems therefore need to be ready to respond to the myriad of challenges following a TSCI by providing access to specialized and comprehensive services. The provision of specialized care in a time-sensitive manner has shown to be crucial for survival and recovery of functioning after a traumatic spinal cord injury (TSCI). However, little is known about the provision of TSCI care in different international contexts; information which is required for strengthening policy and practice.

DETAILED DESCRIPTION:
Like many unforeseen medical emergencies, a TSCI could lead to early death in the absence of essential emergency and acute care. Hence, the single most important indicator of the quality of medical care is reflected in short- and long-term mortality. However, in order to improve survival after TSCI, it is also important to identify factors and processes of routine practice related to mortality. This could be accomplished by examining the extent to which processes of care reflect international guidelines and standards. These guidelines specifically stress the importance of a systematic approach towards the management of TSCI, which include specialized and comprehensive care that is delivered in a multi-disciplinary manner. More specifically, established success factors of TSCI healthcare have proven to include appropriate emergency management (e.g. transfer logistics to trauma unit), early spinal surgery and admission to specialist units, as well as multidisciplinary care. As a collective, literature has shown that a systematic approach towards the management of TSCI leads to a reduction in mortality, secondary complications and re-hospitalizations, as well as better functional outcomes.

In Sweden, a systematic approach towards the management of TSCI was initiated around the 1970's. A number of studies investigating the acute management and mortality after TSCI found better aligned processes of care, and significantly greater survival, in Sweden, compared with a non-systematic approach to care followed in Greece. More specifically, transfer logistics from the accident scene to a specialized trauma unit, key therapeutic interventions, and timing of spinal surgery were better aligned to the international guidelines for the acute management of adults with SCI. In addition, numerous societal services, such as vocational rehabilitation, modifications of living conditions and workplace insurance, are provided to survivors of TSCI to enhance their independence and societal participation.

Unlike Sweden, South Africa had yet to fully implement a systematic healthcare approach to TSCI management. Access to specialized healthcare services is not only a historic problem in South Africa, but it is further exacerbated by the lack of resources. Only one specialized SCI unit is available in South Africa, serving around 8 million people in the Western Cape Province. With the high incidence of TSCI in South Africa, mainly high risk TSCI patients (e.g. those in need of stabilizing spinal surgery) get access to specialized care at the SCI unit. In contrast, those not prioritized for treatment at the specialized SCI unit are treated at hospitals, including both secondary and tertiary level of care, providing non-specialized SCI health care. The common occurrence of non-specialized care of TSCI survivors in South Africa is alarming, especially as such care has shown to be related to a high mortality rate and the occurrence of preventable secondary complications. To improve the outcome of TSCI in South Africa, there is a crucial need to audit the nature and timing of essential processes of care and model their relationship with mortality, complications and long-term outcomes. Furthermore, given the low one-year mortality in Sweden, a comparison of processes of care between Sweden and South Africa could provide empirical evidence pointing to processes which could be modified.

As a first step to strengthening the management guidelines for TSCI care in South Africa, the overarching aim of this study is to explore health-care processes and outcomes of TSCI care in South Africa and Sweden. Specific aims are to: 1) describe acute processes of TSCI care in South Africa and Sweden in comparison to international guidelines, 2) determine acute- and long-term outcomes of TSCI care, including survival status, secondary complications and functioning in South Africa and Sweden and 3) identify predictors for survival, secondary complications and functioning 12 months post-injury in South Africa and Sweden.

ELIGIBILITY:
Inclusion Criteria:

* A TSCI defined as a sudden loss of voluntary muscle strength, sensation and autonomic functions below the level of injury, which will vary depending on neurological level of injury and extent of impairment, but must include altered sacral sensation;
* The injury must result in persisting impairment (i.e. not just a concussion) after emergence from neurogenic shock, which generally occurs within the first 24-72 hours after injury;
* Abnormal imaging, such as with Magnetic Resonance Imaging scan or multi-slice Computed Tomography scan;
* 18 years of age;
* Residents of one of the two study settings;
* Those admitted to the government-funded hospitals providing SCI care;
* Those consenting to participate in the study

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All newly-injured individuals with traumatic spinal cord injury for at least a one-year period within a defined catchment area.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Mortality | at the end of acute hospital care (approximately six weeks from admission)
  To determine the mortality rate at the end of acute care
One-year mortality | one year after injury
  To determine the mortality rate after traumatic spinal cord injury one-year after injury onset
Prevalence of pressure ulcers | acute care prevalence (within a six-week period approximately)
  To determine the prevalence and grade of pressure ulcers during acute care
Prevalence of pressure ulcers | One year after injury onset
  To determine the prevalence of pressure ulcers one-year after injury
Change in neurological classification from baseline to the end of acute care according to the American Spinal Injury Association Impairment Scale | End of acute care (within a six-week period approximately)
  Neurological status using the ASIA scale (A-E)
Change in neurological classification from the end of acute care to one-year after injury according to the American Spinal Injury Association Impairment Scale | One year after injury onset
  Neurological status using the ASIA scale (A-E)

SECONDARY OUTCOMES:
Change in activity limitations from acute care admission to end of acute admission according to the Spinal Cord Independence Measure III | After acute care (approximately 6 weeks post injury)
  Change in activity limitations according to Spinal Cord Independence Measure III
Change in activity limitations from the end of acute care to one-year after injury according to the Spinal Cord Independence Measure III | One-year after injury onset
  Change in activity limitations from the end of acute care (baseline) to one-year after injury according to the Spinal Cord Independence Measure III
Change in health-related quality of life from acute care admission to end of acute care hospitalisation using the EQ-5D measure | At the end of acute care (approximately six weeks)
  Change in health-related quality of life from acute care admission to end of acute care hospitalisation using the EQ-5D measure
Change in health-related quality of life between the end of acute care hospitalisation and one-year after injury onset using the EQ-5D measure | one-year after injury onset
  Change in health-related quality of life between the end of acute care hospitalisation and one-year after injury onset using the EQ-5D measure

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Western Cape, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
May be made available upon reasonable request.